CLINICAL TRIAL: NCT02717455
Title: Phase 1 Trial of Panobinostat in Children With Diffuse Intrinsic Pontine Glioma
Brief Title: Trial of Panobinostat in Children With Diffuse Intrinsic Pontine Glioma
Acronym: PBTC-047
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-047; 5UM1CA081457 (NIH); NCT02899715 (obsolete NCT alias)
Record Dates: First submitted 2016-02-22; First posted 2016-03-23 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Glioma
Keywords: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma; H3K27M; DIPG; DMG
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (STRATUM 1) (Experimental): Patients with recurrent/progressive DIPG will be enrolled at the time of progression. All patients will take the study drug panobinostat (LBH589).
  Interventions: Drug: LBH589
- Treatment (STRATUM 2) (Experimental): Patients with non-progressed DIPG or H3K27M+ Thalamic DMG will be enrolled. All patients will take the study drug panobinostat (LBH589).
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — STRATUM 1: Recurrent/progressive DIPG. Panobinostat will be given every other day, 3 times/ week, p.o. preferably on Mon/Wed/Fri, for three weeks, followed by one week off of therapy. Three weeks of therapy plus the one week rest period (4 weeks) will constitute one course. Treatment will continue for up to 26 courses (about 2 years) barring progressive disease or unacceptable toxicity.
  STRATUM 2: Non-progressed DIPG or H3K27M+ Thalamic DMG. Panobinostat will be given every other day, 3 times/week, every other week p.o. preferably on Mon/Wed/Fri. Four weeks will constitute one course. Treatment will continue for up to 26 courses (about 2 years) unless the patient experiences progressive disease, unacceptable toxicity or any of the off-treatment criteria.
  Other Names: Panobinostat

SUMMARY:
This phase I trial studies the side effects and best dose of panobinostat in treating younger patients with diffuse intrinsic pontine glioma (DIPG). Panobinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Stratum 1 treats patients with DIPG that has returned or gotten worse (progressed). Stratum 2 treats patients with DIPG or H3K27+Thalamic Diffuse Malignant Glioma (DMG) that has not yet gotten worse.

DETAILED DESCRIPTION:
Description

This is a multicenter, phase 1 trial of Panobinostat (LBH589) for children with diffuse intrinsic pontine glioma tumors.

Panobinostat is a pan-HDAC inhibitor of Class I, II and IV histone deacetylases (HDACs) involved in the deacetylation of histone and non-histone cellular proteins. Panobinostat inhibits purified total cellular histone deacetylase activity (IC50 = 0.03 uM) and activities of most HDAC isoforms (IC50 <10nM). In addition, panobinostat induces expression of the cell-cycle control genes including CDKN1A (p21), and selectively inhibits the proliferation of a variety of tumor cells compared to normal cells. It has been extensively profiled for its in vitro and in vivo pharmacological activity on a variety of tumor cell lines and tumor xenograft mice models.

Based on the in vitro and in vivo activity of panobinostat in preclinical models using DIPG cell cultures and orthotopic xenograft model systems, and the potentially important role of histone deacetylases and histone 3 K27M mutations in relation to pontine malignancies, the investigators are conducting a Phase 1 study of panobinostat in children with recurrent/progressive DIPG.

The primary objectives of the study are to (1) describe the toxicity profile and define the dose-limiting toxicities of panobinostat in children with recurrent/progressive DIPG, or with non-progressed DIPG or H3K27+Thalamic Diffuse Malignant Glioma (DMG) taken every other week; (2) estimate the maximum tolerated dose and/or the recommended Phase 2 dose of panobinostat in children with recurrent/progressive DIPG, or with non-progressed DIPG or H3K27+Thalamic Diffuse Malignant Glioma (DMG) taken every other week; and (3) evaluate and characterize the plasma pharmacokinetics of panobinostat in children with recurrent/progressive DIPG, or with non-progressed DIPG or H3K27+Thalamic Diffuse Malignant Glioma (DMG) taken every other week.

Schema

STRATUM 1:

Only patients with recurrent or progressive DIPG will be enrolled initially. Panobinostat will be administered every other day, 3 times/week, p.o. preferably on a Monday/Wednesday/Friday schedule for three weeks, followed by a rest period. Three weeks of therapy plus the one week rest period (total 4 weeks) will constitute one course. Treatment will continue for up to two years (26 courses) unless the patient experiences progressive disease, unacceptable toxicity or any of the off-study criteria.

The starting dose (dose level 1) is 10 mg/m2/day. Below are the proposed dose levels to be studied:

Dose level # Panobinostat oral dose (mg) Minimum BSA Restriction

0*: 5 mg/m2/day MWF, three weeks on, one week off (1 course = 28 days). Patients must have a BSA ≥ 0.80 m2.

1 (starting dose level): 10 mg/m2/day MWF, three weeks on, one week off, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

2: 16 mg/m2/day MWF, three weeks on, one week off, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

3: 22 mg/m2/day MWF, three weeks on, one week off, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

4: 28 mg/m2/day MWF, three weeks on, one week off, (1 course = 28 days). Patients must have a BSA ≥ 0.50 m2.

5: 36 mg/m2/day MWF, three weeks on, one week off, (1 course = 28 days). Patients must have a BSA ≥ 0.50 m2.

Panobinostat will be administered as a single agent

* Dose level 0 represents a potential treatment dose for patients requiring a dose reduction from dose level 1 and may be used as a contingency dose level if the starting dose level of panobinostat is not tolerated in the initial cohort.

STRATUM 2:

Patients with DIPG or H3K27+Thalamic Diffuse Malignant Glioma (DMG) who have received adequate radiation therapy but have not yet progressed will be enrolled in the currently open Stratum 2. Panobinostat will be administered every other day, 3 times/week, every other week p.o. preferably on a Monday/Wednesday/Friday schedule. Total 4 weeks will constitute one course. Treatment will continue for up to two years (26 courses) unless the patient experiences progressive disease, unacceptable toxicity or any of the off-treatment criteria.

The starting dose (dose level 1) is 16 mg/m2/day. Below are the proposed dose levels to be studied:

Dose level # Panobinostat oral dose (mg) Minimum BSA Restriction

Negative 1*: 5 mg/m2/day MWF, every other week (1 course = 28 days). Patients must have a BSA ≥ 0.80 m2.

0*: 10 mg/m2/day MWF, every other week, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

1 (expected starting dose level): 16 mg/m2/day MWF, every other week, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

2: 22 mg/m2/day MWF, every other week, (1 course = 28 days). Patients must have a BSA ≥ 0.65 m2.

3: 28 mg/m2/day MWF, every other week, (1 course = 28 days). Patients must have a BSA ≥ 0.50 m2.

4: 36 mg/m2/day MWF, every other week, (1 course = 28 days). Patients must have a BSA ≥ 0.50 m2.

Panobinostat will be administered as a single agent

* Dose levels 0 and -1 represent potential treatment doses for patients requiring a dose reduction from dose level 1 and may be used as a contingency dose level if the starting dose level of panobinostat is not tolerated in the initial cohort.

ELIGIBILITY:
STRATUM 1 - INCLUSION CRITERIA

* DIAGNOSIS - Patients with progressive DIPG or H3K27M+ Thalamic DMG , as defined by progressive neurologic abnormalities or worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid toxicity wean, electrolyte disturbances, sepsis, hyperglycemia, etc.), OR an increase in the bi-dimensional measurement, taking as a reference the smallest disease measurement recorded since diagnosis, OR the appearance of a new tumor lesion since diagnosis.

  * Please note: patients with a radiographically typical DIPG, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation.
  * Patients with pontine lesions that do not meet these radiographic criteria will be eligible if there is histologic confirmation of malignant glioma WHO II-IV.
  * Thalamic Diffuse Midline Glioma patients will be eligible if there is tissue confirmation of the H3K27M mutation by immunohistochemistry or by gene testing performed in a CLIA certified laboratory of the investigator's choice.
* AGE - Patients must be ≥ 2 but < 22 years of age at the time of enrollment.
* BSA

  * Patients must have a BSA ≥ 0.80 m2 for dose 5mg/m2.
  * Patients must have a BSA ≥ 0.65 m2 for doses of 10mg/m2 - 22 mg/m2.
  * Patients must have a BSA ≥ 0.50 m2 for doses of 28 mg/m2 - 36 mg/m2.
* ABILITY TO SWALLOW - Patient must be able to swallow capsules whole.
* PERFORMANCE STATUS - Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within 7 days of enrollment must be ≥ 50%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* PRIOR THERAPY - Patients must have received a minimum of 54 Gy focal irradiation administered over approximately 42 days prior to enrollment. Patients must have recovered from the acute treatment-related toxicities (defined as < grade 1) of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* MYELOSUPPRESSIVE CHEMOTHERAPY - Patients must have received their last dose of known myelosuppressive anticancer therapy or immunotherapy at least 21 days prior to enrollment (42 days if prior nitrosourea).
* INVESTIGATIONAL/ BIOLOGIC AGENT:

  * Biologic or investigational agent (anti-neoplastic): Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment. (For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur, and discussed with the principal investigator.)
  * Monoclonal antibody treatment and agents with known prolonged half-lives: At least three half-lives must have elapsed prior to enrollment. (Note: A list of the half-lives of commonly used monoclonal antibodies is available on the PBTC webpage under Generic Forms and Templates.)
* RADIATION THERAPY - Patients must have had their last fraction of:

  * Craniospinal irradiation or radiation to ≥ 50% of pelvis > 3 months prior to enrollment.
  * Focal irradiation to the primary site > 42 days prior to enrollment
  * Local palliative irradiation other than previously irradiated primary site (small port) ≥ 14 days
* ORGAN FUNCTION - Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/mm3
  * Platelets ≥ 100,000/ mm3 (unsupported, defined as no platelet transfusion within 7 days, and recovery from post-transfusion nadir)
  * Hemoglobin ≥ 8 g/dl (may receive transfusions)
  * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
  * ALT(SGPT) < 3 x institutional upper limit of normal
  * Albumin ≥ 3 g/dl
  * Potassium ≥ LLN
  * Serum total calcium (correct for serum albumin) or ionized calcium ≥ LLN
  * Serum creatinine based on age/gender as noted below. Patients that do not meet the criteria below but have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 ml/min/1.73 m2 are eligible. Maximum Serum Creatinine for age/gender:

    * Age 2 to < 6 years: 0.8 mg/dL (male); 0.8 mg/dL (female)
    * Age 6 to < 10 years: 1 mg/dL (male); 1 mg/dL (female)
    * Age 10 to < 13 years: 1.2 mg/dL (male); 1.2 mg/dL (female)
    * Age 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)
    * Age ≥ 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
  * Cardiac Function:

    * Left ventricular ejection fraction ≥ 50 by gated radionuclide study OR shortening fraction of ≥ 27% by echocardiogram
    * Patient has no ventricular arrhythmias except for benign premature ventricular contractions.
    * Patient has a QTc interval < 450 ms.
* GROWTH FACTORS - Patients must be off all colony-forming growth factor(s) for at least 7 days prior to enrollment (i.e. filgrastim, sargramostim or erythropoietin). 14 days must have elapsed if patients received PEG formulations.
* FRUIT - Patients must agree to avoid grapefruit or grapefruit juice and Seville (sour) oranges during the entire study.
* PREGNANCY STATUS - Female patients of childbearing potential must have a negative serum or urine pregnancy test.
* PREGNANCY PREVENTION - Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for 3 months after the last dose of panobinostat.
* INFORMED CONSENT - The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.

STRATUM 1 - EXCLUSION CRITERIA

* PRIOR THERAPY

  * Patients who have had > 60 Gy total radiation to the pons (e.g. patients who have received re-irradiation).
  * Patients have had prior HDAC, DAC, HSP90 inhibitors for the treatment of their DIPG.
  * Patients have had valproic acid within 28 days prior to enrollment.
  * Patients have had prior bone marrow transplant.
* NEUROLOGICAL STATUS - Patients have significant acute deterioration in neurologic status in 72 hours prior to enrollment, in the opinion of the treating physician.
* GASTROINTESTINAL

  * Patients have impairment of GI function or GI disease that may significantly alter the absorption of panobinostat; for example severe inflammatory bowel disease.
  * Patients have diarrhea > CTCAE grade 2.
* SYSTEMIC ILLNESS - Patients have any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the ability of the patient to tolerate protocol therapy or put them at additional risk for toxicity or would interfere with the study procedures or results.
* OTHER MALIGNANCY - Patients have a history of any other malignancy.
* TRANSFUSIONS - Patients are known to be refractory to red blood cell or platelet transfusions.
* CONCURRENT THERAPY

  * Patients who are receiving any other anticancer or investigational drug therapy
  * Patients who are required to receive any medication which can prolong the QTc interval. Please see Protocol Appendix B: Medications Which May Cause QTc Prolongation.
* BREASTFEEDING - Female patient IS breastfeeding.
* INABILITY TO PARTICIPATE - Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions

STRATUM 2 - INCLUSION CRITERIA

* DIAGNOSIS - Patients with DIPG who have not yet progressed by clinical or radiographic criteria.

  * Please note: patients with a radiographically typical DIPG, defined as a tumor with a pontine epicenter and diffuse involvement of more than 2/3 of the pons, are eligible without histologic confirmation.
  * Patients with pontine lesions that do not meet these radiographic criteria will be eligible if there is histologic confirmation of malignant glioma WHO II-IV.
* AGE - Patients must be ≥ 2 but < 22 years of age at the time of enrollment.
* BSA Patients must have a BSA ≥ 0.80 m2 for dose 5mg/m2. Patients must have a BSA ≥ 0.65 m2 for doses of 10mg/m2 - 22 mg/m2. Patients must have a BSA ≥ 0.50 m2 for doses of 28 mg/m2 - 36 mg/m2.
* ABILITY TO SWALLOW - Patient must be able to swallow capsules whole.
* PERFORMANCE STATUS - Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within 7 days of enrollment must be ≥ 50%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* PRIOR THERAPY - Patients must have received a minimum of 54 Gy focal irradiation administered over approximately 42 days prior to enrollment. Patients must not have received any other prior therapy for treatment of their CNS malignancy besides standard radiation therapy.

  o Patients must have recovered from the acute treatment-related toxicities (defined as < grade 1) of radiotherapy prior to entering this study.
* RADIATION THERAPY - Patients must have had their last fraction of focal irradiation to the primary site > 14 days prior to enrollment. Patients must not have received local palliative irradiation or craniospinal irradiation.
* ORGAN FUNCTION - Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/mm3
  * Platelets ≥ 100,000/ mm3 (unsupported, defined as no platelet transfusion within 7 days, and recovery from post-transfusion nadir)
  * Hemoglobin ≥ 8 g/dl (may receive transfusions)
  * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN)
  * ALT(SGPT) < 3 x institutional upper limit of normal
  * Albumin ≥ 3 g/dl
  * Potassium ≥ LLN
  * Serum total calcium (correct for serum albumin) or ionized calcium ≥ LLN
  * Serum creatinine based on age/gender as noted below. Patients that do not meet the criteria in Table 9 but have a 24-hour Creatinine Clearance or GFR (radioisotope or iothalamate) ≥ 70 ml/min/1.73 m2 are eligible.

    * Age 2 to < 6 years: 0.8 mg/dL (male); 0.8 mg/dL (female)
    * Age 6 to < 10 years: 1 mg/dL (male); 1 mg/dL (female)
    * Age 10 to < 13 years: 1.2 mg/dL (male); 1.2 mg/dL (female)
    * Age 13 to < 16 years: 1.5 mg/dL (male); 1.4 mg/dL (female)
    * Age ≥ 16 years: 1.7 mg/dL (male); 1.4 mg/dL (female)
* CARDIAC FUNCTION:

  * Left ventricular ejection fraction ≥ 50 by gated radionuclide study OR shortening fraction of ≥ 27% by echocardiogram
  * Patient has no ventricular arrhythmias except for benign premature ventricular contractions.
  * Patient has a QTc interval < 450 ms.
* GROWTH FACTORS - Patients must be off all colony-forming growth factor(s) for at least 7 days prior to enrollment (i.e. filgrastim, sargramostim or erythropoietin). 14 days must have elapsed if patients received PEG formulations.
* FRUIT - Patients must agree to avoid grapefruit or grapefruit juice and Seville (sour) oranges during the entire study.
* PREGNANCY STATUS - Female patients of childbearing potential must have a negative serum or urine pregnancy test.
* PREGNANCY STATUS - Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study and for 3 months after the last dose of panobinostat.
* INFORMED CONSENT - The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines.

STRATUM 2 - EXCLUSION CRITERIA

* PRIOR THERAPY - Patients who have had > 60 Gy total radiation to the pons or thalamus (e.g. patients who have received re-irradiation)
* NEUROLOGICAL STATUS - Patients have significant acute deterioration in neurologic status in 72 hours prior to enrollment, in the opinion of the treating physician.
* GASTROINTESTINAL

  * Patients have impairment of GI function or GI disease that may significantly alter the absorption of panobinostat; for example severe inflammatory bowel disease.
  * Patients have diarrhea > CTCAE grade 2.
* SYSTEMIC ILLNESS - Patients have any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the ability of the patient to tolerate protocol therapy or put them at additional risk for toxicity or would interfere with the study procedures or results.
* OTHER MALIGNANCY - Patients have a history of any other malignancy.
* TRANSFUSIONS - Patients are known to be refractory to red blood cell or platelet transfusions.
* CONCURRENT THERAPY

  * Patients who are receiving any other anticancer or investigational drug therapy
  * Patients who are required to receive any medication which can prolong the QTc interval. Please see Appendix B: Medications Which May Cause QTc Prolongation.
* BREASTFEEDING - Female patient is breastfeeding.
* INABILITY TO PARTICIPATE - Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Monje, MD, Phd, Principal Investigator — Stanford University
Locations (10):
- United States (10):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University and Lucile Packard Children's Hospital, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients between 2 and 22 years of age (>= 2, < 22) at the time of enrollment were enrolled at Pediatric Brain Tumor Consortium (PBTC) member institutions. The first patient on study was enrolled on June 28, 2016, and the last patient was enrolled on November 10, 2021.
Pre-assignment Details: Patients with recurrent/progressive diffuse intrinsic pontine glioma (DIPG) were enrolled on stratum 1, and patients with non-progressed DIPG or H3K27M+ thalamic diffuse malignant glioma (DMG) were enrolled on stratum 2.
Groups:
- Stratum 1, Dose Level 1 (10 mg/m^2): Recurrent or progressive DIPG patients received panobinostat orally every other day, 3 times per week at 10 mg/m^2/day for three weeks on, one week off (1 course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 1, Dose Level 2 (16 mg/m^2): Recurrent or progressive DIPG patients received panobinostat orally every other day, 3 times per week at 16 mg/m^2/day for three weeks on, one week off (1 course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 2, Dose Level 1 (16 mg/m^2): Non-progressed DIPG or H3K27M+ thalamic DMG patients received panobinostat orally every other day, 3 times per week at 16 mg/m^2/day for every other week (1 course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 2, Dose Level 2 (22 mg/m^2): Non-progressed DIPG or H3K27M+ thalamic DMG patients received panobinostat orally every other day, 3 times per week at 22 mg/m^2/day for every other week (1 course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 2, Dose Level 3 (28 mg/m^2): Non-progressed DIPG or H3K27M+ thalamic DMG patients received panobinostat orally every other day, 3 times per week at 28 mg/m^2/day for every other week (1course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 2, Dose Level 4 (36 mg/m^2): Non-progressed DIPG or H3K27M+ thalamic DMG patients received panobinostat orally every other day, 3 times per week at 36 mg/m^2/day for every other week (1course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Started | 13 | 6 | 3 | 12 | 12 | 7
Completed | 10 | 5 | 3 | 6 | 7 | 2
Not Completed | 3 | 1 | 0 | 6 | 5 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 2 | 1
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Did not receive study drug | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Extended delay in start of next cycle for reasons unrelated to treatment | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Patient off-treatment for other complicating disease | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Summary statistics for baseline characteristics are shown for all enrolled patients (n = 53).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2) | Total
Number analyzed (Participants) | 13 | 6 | 3 | 12 | 12 | 7 | 53
Age, Continuous [Median (Full Range); unit: years] | 5.9 [3.2 to 20.8] | 10.5 [6.0 to 21.4] | 13.6 [9.9 to 17.3] | 8.0 [4.1 to 16.7] | 7.8 [4.7 to 9.2] | 6.7 [3.5 to 13.6] | 7.9 [3.2 to 21.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 2 | 8 | 7 | 5 | 35
  Male | 3 | 3 | 1 | 4 | 5 | 2 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 2 | 2 | 4 | 13
  Not Hispanic or Latino | 9 | 3 | 2 | 8 | 7 | 3 | 32
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 3 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 3 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 1 | 0 | 4
  White | 6 | 6 | 2 | 3 | 6 | 7 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 6 | 5 | 0 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as adverse events that were at least possibly related to panobinostat that occurred during the first 4 weeks of therapy regardless of expectedness. Hematologic DLTs included grade 4 thrombocytopenia, grade 3 thrombocytopenia with bleeding, grade 3 thrombocytopenia that occurs twice within a treatment course, myelosuppression that causes greater than a 14-day delay between treatment courses, grade 4 neutropenia, grade 3 or 4 febrile neutropenia. Non-hematologic DLTs included any grade 3 or greater non-hematologic toxicities with a few exclusions (such as grade 3 nausea/vomiting that is responsive to antiemetics and that resolves to grade 2 or lower within 5 days, etc.), any grade 2 non-hematological toxicity that persists for more than 7 days and is considered sufficiently medically significant or sufficiently intolerable by patients, and any panobinostat-related non-hematological toxicity that results in a delay of treatment > 14 days between treatment courses.
Time Frame: 4 weeks
Population: Patients who were evaluable for DLT assessment were included in this analysis. Of all 53 patients enrolled, 7 patients were not evaluable for DLT assessment: 4 patients received less than required dose of study drug, 2 patients did not start protocol therapy, and 1 patient had insufficient labs to monitor for DLTs.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 12 | 5 | 3 | 10 | 11 | 5
Participants | 0 | 2 | 0 | 1 | 4 | 3

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Panobinostat in Stratum 1
Description: The MTD of panobinostat was defined as the dose at which the continual reassessment method (CRM) estimated that 25% of patients were expected to experience DLTs. Stratum 1 consisted of recurrent or progressive diffuse intrinsic pontine glioma (DIPG) patients who were treated with the "3 times/week, three weeks on, one week off" schedule (1 course = 28 days).
Time Frame: 4 weeks
Population: Patients who were enrolled on stratum 1 and were evaluable for dose finding assessment were used to determine the MTD for stratum 1. Of 19 patients enrolled on stratum 1, 2 patients were not evaluable for dose finding assessment due to receiving less than required dose of study drug. The remaining 17 patients were used to determine the MTD for stratum I.
Measure: Number; unit: mg/m^2/day
Groups:
- Stratum 1: Recurrent/progressive DIPG patients who were treated with the "3 times/week, three weeks on, one week off" schedule.
Arm/Group | Stratum 1
Number analyzed (Participants) | 17
mg/m^2/day | 10

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Panobinostat in Stratum 2
Description: The MTD of panobinostat was defined as the dose at which the continual reassessment method (CRM) estimated that 25% of patients were expected to experience DLTs. For Stratum 2, non-progressed DIPG or H3K27M+ thalamic diffuse malignant glioma (DMG) patients who completed conventional radiation treatment were eligible. All patients enrolled on this stratum had DIPG tumors and were treated with the "3 times/week, every other week" schedule (1 course = 28 days).
Time Frame: 4 weeks
Population: Patients who were enrolled on stratum 2 and were evaluable for dose finding assessment were used to determine the MTD for stratum 2. Of 34 patients enrolled on stratum 2, 5 patients were not evaluable due to: receiving less than required dose of study drug (2), disease progression before active treatment (1), withdrawal/refusal prior to protocol therapy (1), and insufficient labs to monitor for dose-limiting toxicities (1). The remaining 29 patients were used to determine the MTD for stratum 2.
Measure: Number; unit: mg/m^2/day
Groups:
- Stratum 2: Non-progressed DIPG or H3K27M+ thalamic DMG patients who were treated with the "3 times/week, every other week" schedule.
Arm/Group | Stratum 2
Number analyzed (Participants) | 29
mg/m^2/day | 22

4. Primary Outcome: Volume of Distribution (Vd)
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at pre-dose and at 0.5, 1, 2, 4, 8 (±1), 24 (±4) hours after the first dose of panobinostat, as well as prior to the second dose on Course 1 Day 3. Volume of distribution (Vd) was estimated using a noncompartmental method.
Time Frame: Up to day 3
Population: Patients who had PK samples collected and had Vd data available were included in this analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 10 | 5 | 3 | 7 | 7 | 4
L | 1704 (827) | 2135 (1268) | 3358 (1136) | 2141 (906) | 1967 (455) | 2487 (2760)

5. Primary Outcome: Elimination Rate (Kel)
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at pre-dose and at 0.5, 1, 2, 4, 8 (±1), 24 (±4) hours after the first dose of panobinostat, as well as prior to the second dose on Course 1 Day 3. Elimination rate (Kel) was estimated using a noncompartmental method.
Time Frame: Up to day 3
Population: Patients who had PK samples collected and had Kel data available were included in this analysis.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 10 | 5 | 3 | 7 | 7 | 4
per hour | 0.059 (0.024) | 0.065 (0.013) | 0.047 (0.003) | 0.057 (0.012) | 0.047 (0.006) | 0.066 (0.017)

6. Primary Outcome: Half-life (t1/2)
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at pre-dose and at 0.5, 1, 2, 4, 8 (±1), 24 (±4) hours after the first dose of panobinostat, as well as prior to the second dose on Course 1 Day 3. Half-life (t1/2) was estimated using a noncompartmental method.
Time Frame: Up to day 3
Population: Patients who had PK samples collected and had t1/2 data available were included in this analysis.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 10 | 5 | 3 | 7 | 7 | 4
hour | 13.0 (4.0) | 11.0 (2.0) | 14.7 (1.1) | 12.6 (2.8) | 14.8 (1.9) | 11.3 (3.8)

7. Primary Outcome: Clearance (CL/F)
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at pre-dose and at 0.5, 1, 2, 4, 8 (±1), 24 (±4) hours after the first dose of panobinostat, as well as prior to the second dose on Course 1 Day 3. Clearance (CL/F) was estimated using a noncompartmental method.
Time Frame: Up to day 3
Population: Patients who had PK samples collected and had CL/F data available were included in this analysis.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 10 | 5 | 3 | 7 | 7 | 4
L/h | 87 (19) | 146 (104) | 156 (44) | 115 (34) | 93 (26) | 129 (109)

8. Primary Outcome: Area Under the Curve (AUC)
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at pre-dose and at 0.5, 1, 2, 4, 8 (±1), 24 (±4) hours after the first dose of panobinostat, as well as prior to the second dose on Course 1 Day 3. The area under the curve (AUC) was estimated using a noncompartmental method and calculated from time of dosing to the last measurable concentration.
Time Frame: Up to day 3
Population: Patients who had PK samples collected and had AUC data available were included.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
Number analyzed (Participants) | 12 | 6 | 3 | 10 | 11 | 6
h*ng/mL | 102 (44) | 191 (146) | 143 (64) | 239 (71) | 284 (73) | 372 (222)

9. Secondary Outcome: Progression-free Survival (PFS) in Stratum 1
Description: PFS was measured from the time of treatment initiation until the time of progressive disease (PD) or death due to any cause for patients with an event, or until the time of last follow-up for patients who were progression free.
Time Frame: From date on treatment until date of PD or death due to any cause or date of last follow-up
Population: Recurrent/progressive DIPG patients who were enrolled on stratum 1 and received at least one dose of panobinostat were included in the analysis. Per the associated protocol objective, all dose levels on stratum 1 were combined to estimate the PFS for this stratum.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 1
Number analyzed (Participants) | 19
months | 1.87 [0.73 to 9.00]

10. Secondary Outcome: Overall Survival (OS) in Stratum 1
Description: OS was measured from the time of treatment initiation until the time of death due to any cause for patients who died, or until the time of last follow-up for patients who survived.
Time Frame: From date on treatment until date of death due to any cause or date of last follow-up
Population: Recurrent/progressive DIPG patients who were enrolled on stratum 1 and received at least one dose of panobinostat were included in the analysis. Per the associated protocol objective, all dose levels on stratum 1 were combined to estimate the OS for this stratum.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 1
Number analyzed (Participants) | 19
months | 5.23 [0.73 to 36.60]

11. Secondary Outcome: Progression-free Survival (PFS) in Stratum 2
Description: as for outcome 9
Time Frame: From date on treatment until date of PD or death due to any cause or date of last follow-up
Population: Non-progressed DIPG or H3K27M+ thalamic DMG patients who were enrolled on stratum 2 and received at least one dose of panobinostat were included in the analysis. Per the associated protocol objective, all dose levels on stratum 2 were combined to estimate the PFS for this stratum. Two patients who did not start protocol therapy were excluded.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 2
Number analyzed (Participants) | 32
months | 3.83 [0.23 to 14.93]

12. Secondary Outcome: Overall Survival (OS) in Stratum 2
Description: as for outcome 10
Time Frame: From date on treatment until date of death due to any cause or date of last follow-up
Population: Non-progressed DIPG or H3K27M+ thalamic DMG patients who were enrolled on stratum 2 and received at least one dose of panobinostat were included in the analysis. Per the associated protocol objective, all dose levels on stratum 2 were combined to estimate the OS for this stratum. Two patients who did not start protocol therapy were excluded.
Measure: Median (Full Range); unit: months
Arm/Group | Stratum 2
Number analyzed (Participants) | 32
months | 9.13 [0.23 to 20.30]

13. Secondary Outcome: Percentage of Patients With H3F3A K27M Mutation Detected in Blood Samples
Description: Cell-free DNA based assay was used to determine whether H3F3A K27M mutation could be detected in patients' blood samples. Percentage of patients in whom this mutation was detected was summarized within each stratum and at each time point.
Time Frame: Blood samples were collected for cell-free DNA based assay at Course 1 Day 1 (C1D1), C2D1, C4D1, and C6D1.
Population: Only patients with cell-free DNA assay results available from blood samples were included in this analysis. Per the statistical section in the protocol, percentage of patients in whom the mutation was detected was summarized within each stratum and at each time point.
Measure: Number; unit: Percentage of participants
Groups:
- Stratum 1: Recurrent or progressive DIPG patients who were treated with the "3 times/week, three weeks on, one week off" schedule
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 15 | 18
Percentage of participants
  Course 1 Day 1: number analyzed (Participants) | 15 | 17
  Course 1 Day 1 | 0 | 5.9
  Course 2 Day 1: number analyzed (Participants) | 11 | 13
  Course 2 Day 1 | 0 | 23.1
  Course 4 Day 1: number analyzed (Participants) | 4 | 8
  Course 4 Day 1 | 25.0 | 0
  Course 6 Day 1: number analyzed (Participants) | 0 | 5
  Course 6 Day 1 |  | 20.0

14. Secondary Outcome: Percentage of Patients With Hist1H3B K27M Mutation Detected in Blood Samples
Description: Cell-free DNA based assay was used to determine whether Hist1H3B K27M mutation could be detected in patients' blood samples. Percentage of patients in whom this mutation was detected was summarized within each stratum and at each time point.
Time Frame: Blood samples were collected for cell-free DNA based assay at Course 1 Day 1 (C1D1), C2D1, C4D1, and C6D1.
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 15 | 18
Percentage of participants
  Course 1 Day 1: number analyzed (Participants) | 15 | 17
  Course 1 Day 1 | 0 | 0
  Course 2 Day 1: number analyzed (Participants) | 11 | 13
  Course 2 Day 1 | 0 | 0
  Course 4 Day 1: number analyzed (Participants) | 4 | 8
  Course 4 Day 1 | 0 | 0
  Course 6 Day 1: number analyzed (Participants) | 0 | 5
  Course 6 Day 1 |  | 0

15. Secondary Outcome: Percentage of Patients With H3F3A K27M Mutation Detected in Urine Samples
Description: Per protocol, cell-free DNA based assay was to be used to determine whether H3F3A K27M mutation could be detected in patients' urine samples, and percentage of patients in whom this mutation was detected would be summarized within each stratum and at each time point. With current technologies available to the lab, no patients had cell-free DNA assay results from urine samples.
Time Frame: Urine samples were collected for cell-free DNA based assay at Course 1 Day 1 (C1D1), C2D1, C4D1, and C6D1.
Reporting Status: Not Posted

16. Secondary Outcome: Percentage of Patients With Hist1H3B K27M Mutation Detected in Urine Samples
Description: Per protocol, cell-free DNA based assay was to be used to determine whether Hist1H3B K27M mutation could be detected in patients' urine samples, and percentage of patients in whom this mutation was detected would be summarized within each stratum and at each time point. With current technologies available to the lab, no patients had cell-free DNA assay results from urine samples.
Time Frame: Urine samples were collected for cell-free DNA based assay at Course 1 Day 1 (C1D1), C2D1, C4D1, and C6D1.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 2 years after initiation of protocol treatment
Description: Adverse events (AEs) were graded using CTCAE v4.0. AEs collected per protocol included a) grade 1 or 2 AEs if attribution was at least possibly related to panobinostat, and b) all grade 3+ AEs on treatment and within 30 days off treatment. All these AEs were summarized in SAE and Other AE tables below. All mortalities on this study were due to disease, except one for upper airway obstruction. Two patients on stratum 2 did not start protocol therapy and were not counted as at risk.
Arm/Group | Stratum 1, Dose Level 1 (10 mg/m^2) | Stratum 1, Dose Level 2 (16 mg/m^2) | Stratum 2, Dose Level 1 (16 mg/m^2) | Stratum 2, Dose Level 2 (22 mg/m^2) | Stratum 2, Dose Level 3 (28 mg/m^2) | Stratum 2, Dose Level 4 (36 mg/m^2)
All-Cause Mortality (participants affected / at risk) | 13/13 | 5/6 | 3/3 | 5/11 | 11/12 | 5/6
Serious Adverse Events (participants affected / at risk) | 9/13 | 4/6 | 0/3 | 5/11 | 4/12 | 4/6
Other Adverse Events (participants affected / at risk) | 13/13 | 6/6 | 3/3 | 11/11 | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1, Dose Level 1 (10 mg/m^2) (N=13) | Stratum 1, Dose Level 2 (16 mg/m^2) (N=6) | Stratum 2, Dose Level 1 (16 mg/m^2) (N=3) | Stratum 2, Dose Level 2 (22 mg/m^2) (N=11) | Stratum 2, Dose Level 3 (28 mg/m^2) (N=12) | Stratum 2, Dose Level 4 (36 mg/m^2) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Nervous system disorders - other, specify (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1, Dose Level 1 (10 mg/m^2) (N=13) | Stratum 1, Dose Level 2 (16 mg/m^2) (N=6) | Stratum 2, Dose Level 1 (16 mg/m^2) (N=3) | Stratum 2, Dose Level 2 (22 mg/m^2) (N=11) | Stratum 2, Dose Level 3 (28 mg/m^2) (N=12) | Stratum 2, Dose Level 4 (36 mg/m^2) (N=6)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (6) | 7 (16) | 3 (7)
Cardiac disorders - other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (3) | 2 (3) | 1 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 8 (13) | 9 (15) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (5) | 3 (11) | 5 (7) | 7 (11) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (4) | 2 (2) | 2 (8) | 8 (21) | 8 (23) | 5 (7)
Fatigue (General disorders) | 5 (7) | 3 (3) | 2 (3) | 5 (7) | 5 (6) | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (10) | 2 (3) | 0 (0) | 4 (4) | 1 (2) | 2 (5)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 3 (4) | 0 (0) | 4 (4) | 2 (2) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (2) | 0 (0) | 1 (4) | 2 (2) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 2 (2)
Electrocardiogram qt corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Hemoglobin increased (Investigations) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - other, specify (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 7 (17) | 6 (7) | 0 (0) | 8 (22) | 10 (30) | 4 (19)
Neutrophil count decreased (Investigations) | 2 (2) | 3 (4) | 2 (2) | 5 (13) | 7 (30) | 6 (18)
Platelet count decreased (Investigations) | 10 (14) | 5 (6) | 3 (6) | 10 (21) | 11 (24) | 4 (8)
Weight loss (Investigations) | 0 (0) | 1 (1) | 2 (5) | 2 (2) | 3 (4) | 0 (0)
White blood cell decreased (Investigations) | 4 (4) | 5 (5) | 2 (2) | 8 (24) | 11 (46) | 5 (18)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (3) | 3 (4) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0) | 6 (6) | 5 (6) | 2 (3)
Metabolism and nutrition disorders - other, specify (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02717455/Prot_SAP_000.pdf